CLINICAL TRIAL: NCT00643487
Title: In Vivo Arthroscopic Behavior of the Infrapatellar Plica of the Knee
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Thomas Smallman, Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: Infrapatellar Plica
Record Dates: First submitted 2008-03-04; First posted 2008-03-26 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: Knee physiology; Anterior compartment knee; Infrapatellar plica; Ligamentum mucosum; Enthesis organ; Fat pad of the knee; Patellofemoral kinematics
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: observation of the behavior of the infrapatellar plica
  Interventions: Procedure: observation of the behavior of the infrapatellar plica

INTERVENTIONS:
Procedure: observation of the behavior of the infrapatellar plica — Local anesthesia using bupivicaine will be initiated. The IPP, if present will be injected with contrast material. In order to minimize discomfort, lidocaine 1%, in as small a volume as possible, will be injected into the fat pad under direct vision to avoid any intra-articular damage from the #25 needle. Radiographic visualization will be verified and the knee taken through a full range of passive and active exercises. Active quadriceps contraction in the subject will be performed at 0, 15, 30 60 and 90 degrees of flexion. In so far as is technically possible, the behavior of the IPP will be videotaped and recorded on lateral fluoroscopy.
  Other Names: Knee surgery

SUMMARY:
Anterior knee pain has been an enigmatic problem for orthopedic surgeons. Recent studies, as well as the clinical observation of the principle investigator have suggested that arthroscopic resection of the infrapatellar plica (IPP), a vestigial remnant from embryonic development of no known clinical or biological significance, may eliminate this pain. The mechanism whereby this pain is related to the IPP is unclear. This study will document the mechanical behavior of the IPP, its kinematics, as recorded on video among a group of subjects who are undergoing arthroscopy. Radiographic visualization of the observed behavior will be obtained by injection of contrast material, and then fluoroscopic recording of a standard series of motions. The plica will then be resected to avoid any possibility of residual symptoms related to its presence. Further fluoroscopy of the knee without plical attachment, will allow the kinematic behavior to be assessed. The procedure will then be terminated.

DETAILED DESCRIPTION:
The infrapatellar plica (IPP) of the human knee is vestigial remnant of the embryologic division between the medial and lateral compartments of the knee, present in 85.5% of knees1, felt by some to be of no clinical significance other than acting as a block to visualization an movement during arthroscopy.2 S.J. Kim 3,4, C.R. Boyd 5, and B. Demirag 2006 have documented successful relier of anterior knee pain after resection of the IPP. This study seeks to assess the relationship between knee motion, activation of the extensor apparatus, and the IPP, in essence, the kinematics of the contents of the anterior compartment of the knee. The hypothesis to be evaluated is:

the infrapatellar plica is a structure of fundamental biomechanical significance, allowing the transmission of force from the extensor apparatus to the distal femur through the fat pad, and acting as a restraint and a modulator of fad pad mobility.

Subjects will be identified by the PI at their office visit. The subject will be consented. The consent will be discussed and verified in a second office visit before surgery. The subject will undergo arthroscopy specifically directed toward identifying and treating known pathology. Once this is finished, if an IPP is present, it will be injected with radiographic contrast material. A series of maneuvers will be performed involving passive and active motion of the knee and active contraction of the quadriceps apparatus. Videotape recording and fluoroscopy will be undertaken. The plica will be removed. Another fluoroscopy will be performed. The patient will be followed according to the standard practice for arthroscopy and the defined pathology.

ELIGIBILITY:
must be Healthy subject must be >18 years of age, skeletally mature must bePending knee joint arthroscopy.

may not have Active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion:
  Healthy subject >18 years of age, skeletally mature Pending knee joint arthroscopy.
  Exclusion:
  Active infection
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas V Smallman, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Kim SJ, Min BH, Kim HK. Arthroscopic anatomy of the infrapatellar plica. Arthroscopy. 1996 Oct;12(5):561-4. doi: 10.1016/s0749-8063(96)90195-4. PMID 8902130
- [Background] Kim SJ, Choe WS. Pathological infrapatellar plica: a report of two cases and literature review. Arthroscopy. 1996 Apr;12(2):236-9. doi: 10.1016/s0749-8063(96)90019-5. PMID 8777004
- [Background] Boyd CR, Eakin C, Matheson GO. Infrapatellar plica as a cause of anterior knee pain. Clin J Sport Med. 2005 Mar;15(2):98-103. doi: 10.1097/01.jsm.0000152706.43395.68. PMID 15782055
- [Background] Demirag B, Ozturk C, Karakayali M. Symptomatic infrapatellar plica. Knee Surg Sports Traumatol Arthrosc. 2006 Feb;14(2):156-60. doi: 10.1007/s00167-005-0643-8. Epub 2005 Jul 30. PMID 16059707

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: In order to attempt observation of the behavior of the infrapatellar plica the following protocol was followed: Local anesthesia using bupivicaine was initiated for intra-articular anaesthesia; 1% lidocaine was used for the portals. The IPP, if present will be injected with contrast material. In order to minimize discomfort, lidocaine 1%, in as small a volume as possible, was injected into the fat pad under direct vision to avoid any intra-articular damage from the #25 needle. Radiographic visualization was verified and the knee was taken through a full range of passive and active exercises. Active quadriceps contraction in the subject was performed at 0, 15, 30 60 and 90 degrees of flexion. In so far as is technically possible, the behavior of the IPP was videotaped and recorded on lateral fluoroscopy. The patients underwent completion of the planned procedure, and the normal post-operative course was followed.
Period: Overall Study
Arm/Group | All Participants
Started | 8
Completed | 5
Not Completed | 3
Not completed — Technical difficulty | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants: No new arms or groups were associated with this observational study
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Recording.
Description: Observe the behavior of the IPP of the knee by fluoroscopy. A complete recording was obtained in 2 patients: this implied that the plica,central body, and fat pad were visualized. The patients then completed a series of manouevres which demonstrated the mechanical behavior of the infrapatellar plica-fat pad complex.
Time Frame: During procedure, on average one hour.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 8
Participants
  Complete Recording | 2
  Partial Recording | 3

ADVERSE EVENTS:
Time Frame: On average less than a year.
Groups:
- All Participants: observation of the behavior of the infrapatellar plica: Local anesthesia using bupivicaine will be initiated. The IPP, if present will be injected with contrast material. In order to minimize discomfort, lidocaine 1%, in as small a volume as possible, will be injected into the fat pad under direct vision to avoid any intra-articular damage from the #25 needle. Radiographic visualization will be verified and the knee taken through a full range of passive and active exercises. Active quadriceps contraction in the subject will be performed at 0, 15, 30 60 and 90 degrees of flexion. In so far as is technically possible, the behavior of the IPP will be videotaped and recorded on lateral fluoroscopy.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
It is difficult technically to place percutaneously an 18 gauge spinal needle in the central body of the fat pad in an awake patient who is lightly sedated. We were fortunate to achieve complete films in 2 patients, and partial films in 3 others.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes